CLINICAL TRIAL: NCT04680910
Title: Precision Targeting of Propofol-induced Electroencephalographic Slow Waves: a Novel Phase I Paradigm for Treatment-resistant Major Depressive Disorder
Brief Title: Slow Wave Induction by Propofol to Eliminate Depression (SWIPED) I
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ben J.A. Palanca, Associate Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202008037; U01MH128483 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Treatment-resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Propofol; Anesthetics; Electroencephalography

STUDY DESIGN:
Intervention Model Description: Pilot Study for safety and feasibility (open label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Propofol infusion (Experimental): Serial propofol infusions to maximally and safely induce unconsciousness and EEG slow waves while minimizing burst suppression.
  Interventions: Drug: Propofol; Diagnostic Test: Electroencephalography (EEG); Diagnostic Test: Slow-Wave Activity

INTERVENTIONS:
Drug: Propofol — Targeted propofol infusion in TRD patients will induce sedation with maximal expression of EEG slow waves and minimal burst suppression.
  Other Names: anesthetic
Diagnostic Test: Electroencephalography (EEG) — EEG will be recorded during propofol infusion and during overnight sleep. Sleep EEG data will be acquired for a minimum of one night prior to the first sedation session, providing a baseline measure. Additional overnight sleep recordings will be performed on day of sedation and subsequent nights.
Diagnostic Test: Slow-Wave Activity — Duration of slow waves during sedation will be evaluated using automated approaches. SWA during sedation will be calculated as the total power in the 0.5-4 Hz frequency band/total time in minutes. SWA during N2/N3 sleep will be calculated as the total power in the 0.5-4 Hz frequency band/total time in minutes in the N2 and N3 sleep stages. Delta sleep ratio will be computed from the SWA measured during the first and second N2/N3 cycles.

SUMMARY:
Our hypothesis is that targeted propofol infusion in treatment-resistant depressed patients will induce slow wave activity during sedation and augment subsequent sleep slow wave activity. We will recruit 15 participants for this open label single arm Phase I trial. All participants will undergo two propofol infusions 2-6 days apart, with each infusion maximizing expression of EEG slow waves. To minimize bias, there will be no specific gender or ethnic background consideration for enrollment. This will be a single site investigation at Washington University Medical Center.

DETAILED DESCRIPTION:
Treatment-resistant depression (TRD) in older adults is a leading cause of disability, excess mortality from suicide, and dementia. Cognitive problems and sleep disturbances are common, contributing to recurrence and poor long-term outcomes. Disrupted slow wave sleep is at the nexus of depression and cognitive dysfunction in older adults. Novel approaches to target this core pathophysiology are lacking. Our mechanistic project is designed to elucidate the relationships between TRD and sleep disturbances in older adults. Through personalized infusions targeting electroencephalographic (EEG) patterns, we aim for a systematic characterization of the relationships between the propofol-induced EEG slow waves and enhancement of slow wave sleep. Through the repurposing of propofol as a therapeutic probe, this innovative proposal will establish whether EEG slow waves are a viable therapeutic target for novel antidepressant approaches.

Study Intervention

Propofol will be infused through a peripheral IV, with the assistance of target-controlled infusion software and pumps, with an anticipated infusion duration of 1-2 hours. Concurrent high-density EEG will be acquired, but with an updated recording rig and sensor nets that use either Elefix conductive gel or salt solution. An Axis P3364LV network camera, synchronized to EEG recordings, will provide video for post-hoc analysis. Participants will be discharged home after nurse monitoring and fulfillment of post-anesthetic care unit criteria.

Patients will be instructed by staff on operation of the Dreem headband for at-home overnight sleep EEG recordings. Patients will demonstrate ability to successfully wear the Dreem and initiate recordings without assistance. The device, charger, instruction sheet, and a link to a 2-minute instructional video will be provided to patients. This paradigm has been successful in the acquisition of preoperative sleep recordings in over 150 geriatric cardiac surgical patients and eight patients who underwent ECT for TRD (ClinicalTrials.gov NCT04451135).

Dreem recordings will be obtained prior to the first propofol infusion and on evenings of propofol infusions. Additionally, recordings will be obtained for up to 6 nights within a 2-week period after the final infusion, to evaluate persistence of restoration of sleep architecture. Participants will exchange the device with staff during each in-person visit, to allow device examination and data download.

Planned subgroup analyses include stratification by sex and age. For the purposes of Phase II of the study, additional subgroup analyses will be performed based on baseline sleep structure (e.g. total sleep time and proportion of time in N3 sleep), and time interval separating the two infusions.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 60 or greater
* English speaking (as an interpreter will not be readily available should a participant need to convey any safety concerns during the propofol infusion sessions or require guidance on conducting at-home sleep recordings)
* Treatment-resistant Depression (non-responsive to at least two adequate trials of oral antidepressants for current episode).

Exclusion Criteria:

* Presence of symptomatic coronary artery disease
* Presence of marked congestive heart failure/cardiomyopathy (NYHA > Class III, LVEF <40%, greater than mild RV systolic dysfunction)
* Prior reaction to propofol
* Resting heart rate < 50 bpm
* Treatment with Electroconvulsive therapy/Transcranial Magnetic Stimulation/vagal nerve stimulation within 6 weeks
* Body mass index > 35
* C-SSRS of 4 or greater (active suicidal ideation with some intent and with/without a specific plan)
* MoCA score < 23 (at least mild dementia)
* Non-prescribed used of amphetamines, opioids, marijuana, cocaine, or phencyclidine
* Intake of > 14 beers/week (or equivalent)
* Anesthetic exposure in the past 4 weeks
* Concurrent use of benzodiazepines > 2 mg/day lorazepam or equivalent, trazodone > 50 mg/day, or gabapentin > 600 mg/day.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Propofol Infusion | Up to one week after propofol infusions
  Adverse events and serious adverse events, including incidence, severity, and likelihood of relation to intervention.
  Evaluate whether serial propofol infusions are safe (<5% serious adverse events directly attributable to infusions)
Feasibility of Propofol Infusion - Propofol SWA | During two-hour propofol infusions
  Evaluate in geriatric TRD patients that propofol infusions can efficiently induce EEG slow waves during infusion (SWA for most of the sedation time)
  Sedation slow wave activity (SWA, EEG power within 0.5-4 Hz frequency band) during propofol sedation.
Feasibility of Propofol Infusion - Sleep SWA | Over three-week period of pre- and post- infusion sleep recordings
  Evaluate Change in sleep slow wave activity during N2/N3 Sleep (post-infusion - pre-infusion) Evaluate whether propofol can augment total sleep SWA in greater or equal to 40% of study completers.

SECONDARY OUTCOMES:
Affects on suicidality | Up to 10 weeks after second infusion
  Evaluate whether propofol infusions are associated with augmented suicidality Change in Suicidality (C-SSRS) Suicidality screening for need of emergency psychiatric care.
Affects sleep structure | Over 3-week period of pre- and post- infusion sleep recordings
  Evaluate changes in sleep structure Changes in duration of N3 and REM sleep and proportion of total sleep time for these stages. Delta sleep ratio (DSR, calculated as the SWA of the 1st NREM cycle divided by the SWA of the 2nd NREM cycle). Established markers for sleep macrostructure.
Affects on cognition (MoCA) | comparison of baseline measure to up to 3 weeks after second infusion
  Evaluate changes in cognitive function Change in Cognitive Performance on the MoCA. Examine potential positive or negative changes cognition that may be associated with propofol infusion.
Affects on cognition (Fluid Cognition) | comparison of baseline measure to up to 3 weeks after second infusion
  Evaluate feasibility in evaluating changes in cognitive function Change in Cognitive Performance on the NIH Toolbox Cognition Battery Examine potential positive or negative changes cognition that may be associated with propofol infusion.

OTHER OUTCOMES:
Feasibility of acquiring propofol-associated changes in circadian rhythms | Three-week period spanning pre- and post propofol infusions
  Examine feasibility of acquiring propofol-associated changes on circadian rhythms using a sleep diary These measures are important for evaluating feasibility of collection in Phase II.
Feasibility of acquiring propofol-associated changes in anhedonia | Pre-infusion and up to 10 weeks after second infusion
  Examine feasibility of acquiring propofol-associated changes on anhedonia Measure of anhedonia (SHAPS, scale 0-14) This assesses for change in anhedonia after propofol infusions These measures are important for evaluating feasibility of collection in Phase II.
Feasibility of acquiring propofol-associated changes in depression | Pre-infusion and up to 10 weeks after second infusion
  Examine feasibility of acquiring propofol-associated changes on depression symptoms Measure of Depressive Symptoms (MADRS, 0-60) This assesses for changes in depression after propofol infusions These measures are important for evaluating feasibility of collection in Phase II.
Feasibility of acquiring propofol-associated changes in affect | On days of propofol infusions
  Examine feasibility of acquiring propofol-associated changes on affect Measure of affect (feeling scale) This assesses any affect immediately after propofol infusions These measures are important for evaluating feasibility of collection in Phase II.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be released in manuscript form. Outcome data will be uploaded to the NIMH Data Archive on a rolling basis. EEG data will be shared via the National Sleep Research Resource within three years of study completion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within three years of study completion.
Access Criteria: Data use agreements may be required.

REFERENCES:
- [Background] Murphy MJ, Peterson MJ. Sleep Disturbances in Depression. Sleep Med Clin. 2015 Mar;10(1):17-23. doi: 10.1016/j.jsmc.2014.11.009. Epub 2014 Dec 12. PMID 26055669
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Doghramji K, Jangro WC. Adverse Effects of Psychotropic Medications on Sleep. Psychiatr Clin North Am. 2016 Sep;39(3):487-502. doi: 10.1016/j.psc.2016.04.009. Epub 2016 Jun 24. PMID 27514301
- [Derived] Rios RL, Green M, Smith SK, Kafashan M, Ching S, Farber NB, Lin N, Lucey BP, Reynolds CF, Lenze EJ, Palanca BJA; SWIPED Study Team. Propofol enhancement of slow wave sleep to target the nexus of geriatric depression and cognitive dysfunction: protocol for a phase I open label trial. BMJ Open. 2024 May 30;14(5):e087516. doi: 10.1136/bmjopen-2024-087516. PMID 38816055
- [Derived] Rios RL, Kafashan M, Hyche O, Lenard E, Lucey BP, Lenze EJ, Palanca BJA. Targeting Slow Wave Sleep Deficiency in Late-Life Depression: A Case Series With Propofol. Am J Geriatr Psychiatry. 2023 Aug;31(8):643-652. doi: 10.1016/j.jagp.2023.03.009. Epub 2023 Mar 28. PMID 37105885